CLINICAL TRIAL: NCT05070182
Title: Resting Energy Needs in Brain Dead Patients
Brief Title: Resting Energy Needs in Brain Dead Patients (reSting EneRgy nEeds iN brAin DEad Patients)
Acronym: SERENADE
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Papageorgiou General Hospital (Other)
Responsible Party: Principal Investigator, Chrysoula Pourzitaki, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: 3/24-02.05.2018
Record Dates: First submitted 2021-09-17; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Brain Death; Brain Injuries; Brain Edema; Brain Hemorrhage
Keywords: Resting energy expenditure (REE); Brain Death; Brain injuries
MeSH Terms: conditions — Brain Death; Brain Injuries; Brain Edema; Intracranial Hemorrhages | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with brain damage: ICU patients with brain damage (due to cardiac arrest, intracranial hemorrhage or traumatic brain injury). and GCS upon entry <=8.
  All patients will be examined with a transcranial doppler (TCD) and a metabolic computer (for the measurements of REE) After the final diagnosis the patients' characteristics will be compared according to if they were brain dead or not
  Interventions: Diagnostic Test: REE - Resting Energy Expenditure; Diagnostic Test: Transcranial Doppler

INTERVENTIONS:
Diagnostic Test: REE - Resting Energy Expenditure — REEs represent 60-70% of the needs for a sedentary person and 50% of physically active people.
  For the measurement of REE will be used the metabolic computer (Medical Graphics, Ultima CCM, Minneapolis, USA), which with continuous recording of breath-to-breath volume (Vt), respiratory rate (RR) of ventilation per minute volume (MV) ), of inhaled and exhaled gases (O2 and CO2) has the ability to calculate the values of VO2, VCO2 and with the help of equations the values of REE and RQ.
  All patients in the study will be monitored with the metabolic computer. Their measurements will be recorded every day during their stay in the ICU.
Diagnostic Test: Transcranial Doppler — The measurement of flow velocities in the middle cerebral artery will be done with the transcranial Doppler using a low frequency (2 MHz) ultrasound head.
  All patients entering the study will be examined with the TCD every day during their stay in the ICU.

SUMMARY:
The study will examine the resting energy need (REE) in patients suffering from brain damage. For the measurement of REE will be used a metabolic computer (which with continuous recording of breath-to-breath volume (Vt), respiratory rate (RR) of ventilation per minute volume (MV) ), of inhaled and exhaled gases (O2 and CO2) has the ability to calculate the values of VO2, VCO2 and with the help of equations the values of REE and RQ.

DETAILED DESCRIPTION:
This is a retrospective observational study concerning patients suffering from brain damage.

All the patients suffering from brain damage are monitored in order to examine their resting energy needs (REE). For the measurement of REE the metabolic computer (Medical Graphics, Ultima CCM, Minneapolis, USA) is used.

The main purpose of this study is to reveal the (REE) changing in patients with brain death semiology and examine if the REE changes could be related to the outcome of a patient with intracranial pathology. Moreover the study will examine if the changes in REE measurement are related to changes in flow velocities in the midbrain.

Any measurement shall be preceded by calibration of the metabolic computer pneumotachograph with a 3-liter syringe with an acceptable error of less than 9 ml / lit. The metabolic unit is calibrated for VO2 measurements with two calibration cylinders containing 21% and 12% O2 and for VCO2 measurements with calibration gases containing 5% and 0% CO2 respectively.

The measurement of flow velocities in the middle cerebral artery will be done with the transcranial Doppler using a low frequency (2 MHz) ultrasound head After their final diagnosis (brain death or not) the patients' characteristics will be compared according to the categorization as "brain dead" or not.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients entering the ICU
* Age 18-90 years old
* Clinical Diagnosis of brain damage
* GCS <=8

Exclusion Criteria:

* Patients <18 years old and >90 years old,
* Past history CNS disease (alzheimer's disease, multiple sclerosis, brain tumor, aneurysm) in the last 3 years
* Past history of cachexia due to cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, aged 18-90 years old, entering the ICU, having a GCS <=8 before any intervention, having signs of intracranial damage after a traumatic brain injury or a cardiac arrest succesfull rescucitation or a brain hemorrhage due to aneurysm.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
REE changes | Day 0 (upon entry to ICU) up to 30 days
  Changes in REE in patients with brain damage
MCA changes | Day 0 (upon entry to ICU) up to 30 days
  Changes in flow rates in Median Cerebral Artery (MCA) in patients with brain damage
REE and MCA correlation | Day 0 (upon entry to ICU) up to 30 days
  Correlate the REE changes with those in flow rates in MCA

SECONDARY OUTCOMES:
Prognostic value of REE | Day 0 (upon entry to ICU) up to 30 days
  Compare the values of REE upon entry in the ICU in patients with final diagnosis as brain dead or not

CONTACTS AND LOCATIONS:
Overall Officials: Chryssa Pourzitaki, MD, PhD, Principal Investigator — Faculty of Medicine, School of Health Sciences, Aristotle University of Thessaloniki
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Babikian VL, Feldmann E, Wechsler LR, Newell DW, Gomez CR, Bogdahn U, Caplan LR, Spencer MP, Tegeler C, Ringelstein EB, Alexandrov AV. Transcranial Doppler ultrasonography: year 2000 update. J Neuroimaging. 2000 Apr;10(2):101-15. doi: 10.1111/jon2000102101. PMID 10800264
- [Background] Marinoni M, Alari F, Mastronardi V, Peris A, Innocenti P. The relevance of early TCD monitoring in the intensive care units for the confirming of brain death diagnosis. Neurol Sci. 2011 Feb;32(1):73-7. doi: 10.1007/s10072-010-0407-1. Epub 2010 Sep 25. PMID 20872036
- [Background] Zijlstra N, ten Dam SM, Hulshof PJ, Ram C, Hiemstra G, de Roos NM. 24-hour indirect calorimetry in mechanically ventilated critically ill patients. Nutr Clin Pract. 2007 Apr;22(2):250-5. doi: 10.1177/0115426507022002250. PMID 17374800
- [Background] Bitzani M, Matamis D, Nalbandi V, Vakalos A, Karasakalides A, Riggos D. Resting energy expenditure in brain death. Intensive Care Med. 1999 Sep;25(9):970-6. doi: 10.1007/s001340050991. PMID 10501754